CLINICAL TRIAL: NCT06743412
Title: Ascolto Passivo Di Musica Nella Malattia Cerebrovascolare Acuta
Brief Title: Passive Music Listening in Acute Cerebrovascular Disease
Acronym: MUSICSTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, GIACOMO GIACALONE, MD PhD, IRCCS Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSICSTROKE
Record Dates: First submitted 2024-12-04; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-07

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REGULAR MUSIC LISTENING (Experimental): Patients randomized into this arm are provided with tablet and earphones for regular music listening during hospital stay (1 hour per day in average). After discharge, patients are instructed how to continue regular music listening till the follow-up visit. Patients are required to maintain a daily music listening diary to be presented at the follow-up visit.
  Interventions: Other: Regular music listening
- NO REGULAR MUSIC LISTENING (No Intervention): Patients randomized into this arm do not receive instrumentation for regular music listening during hospital stay. At discharge, patients in this arm are not required to perform regular music listening.

INTERVENTIONS:
Other: Regular music listening — Regular listening of self-selected music sung in Italian language during the hospital stay and after discharge till the follow-up visit after 3 months.
  Arms: REGULAR MUSIC LISTENING

SUMMARY:
The aim of the study is to investigate whether passive music listening during the acute phase of stroke hospitalization is a feasible and acceptable intervention that can improve the patient's psychophysical well-being, reduce anxiety and depression indicators, and improve the patient's perception of their overall health status. Secondly, the effects during hospitalization on physiological parameters, pain perception, quality of sleep, and the use of sedative, antidepressant, or anxiolytic medications will be evaluated. Finally, it will be assessed whether passive music listening is also associated with an improvement in cognitive functions.

The clinical trial is a prospective, randomized, controlled, open-label, single-center study with parallel cohorts.

Subjects with acute cerebrovascular disease (ischemic stroke, hemorrhagic stroke) hospitalized in the Neurology-Stroke Unit at San Raffaele Hospital in Milan will be recruited.

Enrolled subjects will be randomly assigned to 2 groups:

* Group 1: regular music listening starting since the acute phase of hospitalization (between 24 and 96 hours after symptom onset), continuing post-discharge for a total of 3 months.
* Group 2: no regular music listening.

Measurements of psychophysical well-being, anxiety and depression scales, and cognitive functions will be performed at three different time points (baseline, discharge, and 3 months post-ischemic event during the routine follow-up visit as per standard care).

The primary outcome of the study are:

* To evaluate whether passive music listening during hospitalization is associated with an improvement in anxiety/depression levels as measured by the Hospital Anxiety and Depression Scale (HADS).
* To investigate whether passive music listening during hospitalization is associated with an improvement in the patient's perception of their overall health status as measured by the Italian version of the EQ-VAS (EuroQol Visual Analog Scale).
* To assess the feasibility and acceptability of the intervention by measuring the percentage of patients who refuse to participate in the study and the drop-out rate during the hospitalization phase, the percentage of days with music listening during hospitalization, and the total amount of listening hours; through a feasibility, acceptability, and care appreciation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* time of enrollment greater than 24 hours and less than 4 days from onset of acute cerebrovascular disease
* native Italian speaker
* able to cooperate according to the following criteria:

  * NIHSS stroke severity score at enrollment <10.
  * No impairment in alertness, orientation, or language that would prevent adequate communication (NIHSS score <2 for items 1a, 1b, 1c, 9, 10).
  * No known pre-existing severe or moderate cognitive decline (CDR<2).
* potentially able to continue music listening after discharge.
* papable of giving informed consent for the study.

Exclusion Criteria:

* Deafness and/or significant hearing loss and/or significant visual impairment and/or illiteracy.
* Major psychiatric illness.
* Other conditions that, in the investigator's judgment, would prevent compliance with the protocol during hospitalization or the post-hospitalization phase.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in anxiety/depression levels (HADS score) between baseline and discharge. | Baseline vs. discharge (up to 30 days)
  Hospital Anxiety and Depression Scale (HADS), total score ranges between 0-21, with higher values indicating higher levels of anxiety/depression.
Improvement in the patient's perception of overall health status between baseline and discharge (EQ-VAS). | Baseline vs. discharge (up to 30 days)
  EuroQol-visual analogue scales (EQ-VAS). The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Feasibility and acceptability during hospitalization (Percentage of patients who refuse to participate in the study) | Baseline
  Percentage of patients who refuse to participate in the study
Feasibility and acceptability during hospitalization (percentage of drop-outs). | Baseline-discharge (up to 30 days)
  percentage of drop-outs.
Feasibility and acceptability during hospitalization (percentage of days and total hours of music listening during the hospitalization phase). | Baseline-discharge (up to 30 days)
  percentage of days and total hours of music listening during the hospitalization phase.

SECONDARY OUTCOMES:
Improvement in anxiety/depression levels (HADS score) | 3 months (+/- 1 month) follow-up visit
  Hospital Anxiety and Depression Scale (HADS), total score ranges between 0-21, with higher values indicating higher levels of anxiety/depression.
Improvement in the patient's perception of overall health status (EQ-VAS). | 3 months (+/- 1 month) follow-up visit
  EuroQol-visual analogue scales (EQ-VAS). The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Feasibility and acceptability (percentage of drop-outs). | 3 months (+/- 1 month) follow-up visit
  percentage of drop-outs
Evaluation of cognitive functions through MoCA test | Basline vs. discharge (up to 30 days) vs. 3 months (+/- 1 month) follow-up visit
  MoCA (Montreal Cognitive Assessment or The MoCA Test) is a tool for early detection of mild cognitive impairment; total score ranges between 0 and 30, with lower values indicating increasing cognitive impairment.
Evaluation of cognitive functions through Stroop test | Basline vs. discharge (up to 30 days) vs. 3 months (+/- 1 month) follow-up visit
  The time interference score and the error interference score will be measured; according to normative data, the scores will be converted in equivalent scores from 0 to 4 with lower values indicating higher level of impairment.
Evaluation of cognitive functions through delayed story recall | Basline vs. discharge (up to 30 days) vs. 3 months (+/- 1 month) follow-up visit
  The raw score will be converted, according to normative data, to an equivalent score between 0 and 4 with lower values indicating more impairment.
Patient perception of health status related to mobility, usual activities, anxiety, depression, and pain (EQ-5D-3L Italian version). | Baseline vs. discharge (up to 30 days) vs. 3 months (+/- 1 month) follow-up
  The EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version) is a Patient Reported Outcomes (PRO) which examines five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The questionnaire produces a 5-digit health state profile that represents the level of reported problems on each of the five dimensions of health. EQ-5D 5-digit health state is subsequently converted into a single index value, according to normative, which reflects the health state.
Patient perception of sleep quality (ISI insomnia severity index, Italian version). | Baseline vs. discharge (up to 30 days) vs. 3 months (+/- 1 month) follow-up visit
  The total score ranges from 0 to 28, with higher score indicating greater insomnia severity.
Blood pressure, pre- and post-listening. | hospitalization phase (discharge-baseline, up to 30 days)
  Blood pressure, pre- and post-listening to music. Measure unit: mmHg
Daily average number of administrations of sedatives, anxiolytics, and antidepressants. | hospitalization phase (discharge-baseline, up to 30 days)
Heart rate, pre- and post-listening. | hospitalization phase (discharge-baseline, up to 30 days)
  Heart rate, pre- and post-listening to music. Measure unit: beats/min.
Feasibility and acceptability (percentage of days and total hours of music listening). | 3 months (+/- 1 month) follow-up visit
  percentage of days and total hours of music listening.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy